CLINICAL TRIAL: NCT01528800
Title: Inhibit Progression of Coronary Artery Calcification With Vitamin K in HemoDialysis Patients: The iPACK-HD Study
Brief Title: Vitamin K to Attenuate Coronary Artery Calcification in Hemodialysis Patients
Acronym: iPACK-HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Rachel Holden (Other)
Responsible Party: Sponsor-Investigator, Dr. Rachel Holden, Professor of Medicine Queen's University, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: iPACK-HD
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: End-stage Kidney Disease
Keywords: Vitamin K; Chronic Kidney Disease; Vascular Calcification; Hemodialysis; Coronary Artery Calcification
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Vascular Calcification | interventions — Vitamin K 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Microcrystalline Methylcellulose
  Interventions: Drug: Microcrystalline Methylcellulose
- Vitamin K1 (Active Comparator): Vitamin K1
  Interventions: Drug: Vitamin K1

INTERVENTIONS:
Drug: Vitamin K1 — 10mg orally three times a week for 12 months
  Other Names: Phytonadione; Phylloquinone
  Arms: Vitamin K1
Drug: Microcrystalline Methylcellulose — 10mg orally three times a week for 12 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if vitamin K supplementation three times per week reduces the progression of coronary artery calcification over 12 months in dialysis patients compared to placebo.

DETAILED DESCRIPTION:
At every stage of chronic kidney disease (CKD), the leading cause of mortality is cardiovascular disease. This is due, in part, to vascular calcification (VC) of the coronary arteries. The extent of VC in the coronary arteries of patients with CKD is commonly determined by high resolution CT scan. The total coronary artery calcium (CAC) score, measured in Agatston units (AUs), reflects the calcium burden in the three major coronary arteries and is the current standard for determining extent of vascular calcification in hemodialysis patients. Matrix Gla protein (MGP), a vitamin K dependent protein, is a key inhibitor of vascular calcification and is present in the arterial wall. It is established that MGP becomes up-regulated adjacent to sites of calcification and that vitamin K is critical to its function. Therefore vitamin K status may be critical to the extent of vascular calcification in this patient group. However, to date, no trial has examined whether vitamin K supplementation prevents the progression of coronary artery calcification in patients with kidney failure, a group in which high risk has been established. Therefore, our primary research question is: Does vitamin K supplementation with 10 mg of phylloquinone thrice weekly reduce the progression of coronary artery calcification (as measured by CAC score) over 12 months in prevalent hemodialysis patients with a baseline CAC score of ≥ 30 Agatston Units compared to placebo?

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed informed consent
* ≥18 years of age
* Expected to survive one year
* Have end-stage kidney disease and require hemodialysis
* Have a baseline coronary artery calcification score ≥30 Agatston units (AUs)

Exclusion Criteria:

* Have a medical condition that requires warfarin
* Require hemodialysis for acute kidney injury
* Are Pregnant
* Have other severe co-morbid conditions (e.g. malignancy, disabling stroke) with life expectancy less than one year
* Have undergone coronary artery bypass grafting or have stents placed in their coronary arteries
* Are currently enrolled in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 12 months
  Number of participants recruited per month at each site) and an overall crude average of each site's rate.
Compliance with study medication | 12 months
  Proportion of prescribed doses received.
Dropout rate | 12 months
  Proportion of participants who dropped out from the trial.
Adherence to study protocol | 12 months
  Proportion of participants who adhered to the study protocol.
Rates of eligible patients consented and randomized | 12 months
  Proportion of eligible patients consented and randomized.

SECONDARY OUTCOMES:
Coronary artery calcification (Agatston calcium scores) progression | 12 months
  A)The percent and absolute change of the Agatston calcium scores (CT scan) will be assessed at study exit vs. baseline. Included measures will be: Total CAC, Left Main CAC, Right Coronary Artery CAC, Left Anterior Descending CAC, Circumflex CAC, and Posterior Descending Artery CAC.
  B) The proportion of participants with a 15% or greater increase in Agatston calcium scores will be assessed at study exit vs baseline.
Coronary artery calcification (volume calcium scores) progression | 12 months
  A) The percent and absolute change of the volume calcium scores (CT scan) will be assessed at study exit vs. baseline. Included measures will be: Total CAC, Left Main CAC, Right Coronary Artery CAC, Left Anterior Descending CAC, Circumflex CAC, and Posterior Descending Artery CAC.
  B) The proportion of participants with a 15% or greater increase in volume calcium scores will be assessed at study exit vs baseline.
Coronary artery calcification (Agatston calcium scores) regression | 12 months
  The proportion of participants with a 10% or greater decrease in Agatston calcium scores will be assessed at study exit vs baseline.
Coronary artery calcification (volume calcium scores) regression | 12 months
  The proportion of participants with a 10% or greater decrease in volume calcium scores will be assessed at study exit vs baseline.
Aortic valve calcification (Agatston calcium scores) progression | 12 months
  The absolute and percentage change of the Agatston calcium scores (CT scan) will be assessed at study exit vs. baseline.
Aortic valve calcification (volume calcium scores) progression | 12 months
  The absolute and percentage change of the volume calcium scores (CT scan) will be assessed at study exit vs. baseline.
Mitral valve calcification (Agatston calcium scores) progression | 12 months
  The absolute and percentage change of the Agatston calcium scores (CT scan) will be assessed at study exit vs. baseline.
Mitral valve calcification (volume calcium scores) progression | 12 months
  The absolute and percentage change of the volume calcium scores (CT scan) will be assessed at study exit vs. baseline.
Abdominal aortic calcification (AAC) scores | 12 months
  The AAC score (mean score in L1-L4, mean number of positive segments, mean total severity using lateral lumbar spine radiographs) will be assessed at study exit vs. baseline.
Levels of biomarkers of vitamin K status | 12 months
  Gas6, PK, MK4, osteocalcin Gla, osteocalcin Glu, osteocalcin Gla to Glu ratio, percent of osteocalcin undercarboxylated, and dpucMGP will be assessed at baseline, four, eight and study exit. Protein induced by vitamin K absence or antagonist II (PIVKA-II) will be assessed at baseline and study exit.
Prevalence and incidence of thoracic vertebral fractures | 12 months
  The prevalence and incidence of thoracic vertebral fractures (anterior and lateral radiographs) will be assessed at baseline and study exit.
Prevalence and incidence of lumbar vertebral fractures | 12 months
  The prevalence and incidence of lumbar vertebral fractures (anterior and lateral radiographs) will be assessed at baseline and study exit.
Presence/absence and total hospitalizations | 12 months
  The presence or absence and total hospitalizations will be assessed across the study duration per patient.
Presence/absence and total cardiovascular events | 12 months
  The presence or absence and total cardiovascular events (acute coronary syndrome, congestive heart failure, stroke, transient ischemic attack, amputation, and cardiac [symptom-driven] [cerebral or peripheral] revascularization procedure, or cardiac arrest) will be assessed across the study duration per patient.
Presence/absence and total thrombotic events | 12 months
  The presence or absence and total thrombotic events (deep vein thrombosis and pulmonary embolism) will be assessed across the study duration per patient.
Presence/absence and total hemodialysis access thrombotic events | 12 months
  The presence or absence and total hemodialysis access thrombotic events (fistula and/or graft thrombosis or dialysis catheter thrombosis) will be assessed across the study duration per patient.
Presence/absence and total mortality | 12 months
  The presence or absence and total all-cause and cardiovascular cause mortality will be assessed across the study duration per patient.

OTHER OUTCOMES:
Levels of biomarkers of inflammation | 12 months
  C-reactive protein (CRP), interleukin 6 (IL-6), leptin, insulin, glucose, homeostasis model assessment-insulin resistance (HOMA-IR) will be assessed at baseline, four months, eight months, and study exit.
Levels of clinical lab values | 12 months
  Hemoglobin, albumin, Kt/V, creatinine, lipid profile (HDL, LDL, triglycerides, and total cholesterol), and parameters of mineral metabolism (phosphate, calcium, PTH, and ALP) will be assessed monthly. Serum FGF-23 will be assessed at baseline, four months, eight, and study exit.
Concomitant medication assessment (presence/absence/dosage) | 12 months
  Prescription of concomitant medications (listed below) will be assessed monthly.
  * Calcium-based phosphate binders
  * Non-calcium-based phosphate binders
  * Calcitriol
  * Vitamin D Calcimimetic
  * HMG-CoA reductase inhibitors
  * Angiotensin converting enzyme inhibitors
  * Angiotensin II receptor blockers
  * Anti-platelet therapy: acetylsalicylic acid, clopidogrel bisulfate, and dipyridamole
  Average dosage and total exposure across study exit will be assessed for calcitriol, other vitamin D drugs, and calcium-based phosphate binders.
Changes in body composition measures | 12 months
  Muscle atrophy and adipose tissue will be assessed using an L3 slice (CT scan) at study exit vs. baseline. Specifically, muscle, normalized muscle, intermuscular adipose tissue (IMAT), visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT) and total adipose tissue (TAT) cross-sectional area (cm2 or cm2/m2) and muscle, IMAT, VAT and SAT radiodensity (HUs) measurements will be included.
Levels of vascular inflammation variables | 12 months
  Myoglobin, calciprotectin, neutrophil gelatinase-associated lipocalin, matrix-metalloproteinase 2, osteopontin, myeloperoxidase, serum amyloid A, insulin-like growth factor binding protein-4, intercellular adhesion molecule 1, vascular cell adhesion protein 1, matrix-metalloproteinase 9, and cystatin C will be assessed at baseline, four months, eight months and study exit.
Levels of vitamin D metabolites | 12 months
  1,25-OH-D3, 25-OH-D2, percent 25D that is D2, Total 25D, 24,25(OH)2D3, 25D3:24,25D3, 24,25D3:25D3, 3epi25-OH-D3, 3epi25-OH-D3(%), 1,25(OH)2D3, 1,24,25(OH)3D3, 1,25(OH)2D3:1,24,25(OH)3D3, 1,25(OH)2D3:1,24,25(OH)3D3 will be assessed at baseline, four months, eight months and study exit.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Holden, Principal Investigator — Queens University/Kingston Health Sciences Centre: Kingston General Hospital
Locations (3):
- Canada (3):
  - Kingston Health Sciences Centre: Kingston General Hospital Site, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

REFERENCES:
- [Derived] Holden RM, Booth SL, Zimmerman D, Moist L, Norman PA, Day AG, Menard A, Fu X, Shea MK, Babiolakis CS, Nolan R, Turner ME, Ward E, Kaufmann M, Adams MA, Heyland DK. Inhibit progression of coronary artery calcification with vitamin K in hemodialysis patients (the iPACK-HD study): a randomized, placebo-controlled multi-center, pilot trial. Nephrol Dial Transplant. 2023 Feb 28;38(3):746-756. doi: 10.1093/ndt/gfac191. PMID 35641194
- [Derived] Holden RM, Booth SL, Day AG, Clase CM, Zimmerman D, Moist L, Shea MK, McCabe KM, Jamal SA, Tobe S, Weinstein J, Madhumathi R, Adams MA, Heyland DK. Inhibiting the progression of arterial calcification with vitamin K in HemoDialysis patients (iPACK-HD) trial: rationale and study design for a randomized trial of vitamin K in patients with end stage kidney disease. Can J Kidney Health Dis. 2015 May 1;2:17. doi: 10.1186/s40697-015-0053-x. eCollection 2015. PMID 26075081

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT01528800/SAP_000.pdf